CLINICAL TRIAL: NCT00164580
Title: Prevention of HIV Infection in Youth at Risk: Developing Community-Level Intervention Strategies That Work (Community Intervention Trial for Youth (CITY) Study)
Brief Title: Community Intervention Trial for Youth (CITY) Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-1733; U62/CCU113642; U62/CCU513631; U62/CCU513650; U62/CCU513661; U62/CCU913658
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: HIV Infections
Keywords: Homosexuality, Male; Adolescents; Minority Groups; Community Participation; Community Surveys; HIV Seronegativity; HIV
MeSH Terms: conditions — HIV Infections; Homosexuality, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Community-Level Intervention

SUMMARY:
The purpose of this study is to test whether a multi-component, community-level, HIV-prevention intervention is more effective than existing HIV prevention activities in reducing unprotected anal intercourse (UAI) among men ages 15-25 who have sex with men.

DETAILED DESCRIPTION:
In recent years, there have been increases in the rates of unprotected anal intercourse (UAI) reported by men who have sex with men (MSM) and in the numbers of newly diagnosed HIV infections among MSM. Surveys of young MSM (ages 15-29) in numerous U.S. cities from 1994-2000 found an HIV prevalence of 2.2% to 18%, however, HIV prevalence was higher among young MSM of color than among white men. In a survey of 23-29 year-old MSM,nearly 1/3 of African-American men and 15% of Hispanic/Latino men were infected with HIV.

The Community Intervention Trial for Youth (CITY) study is a 13-community randomized control trial designed to evaluate a multi-component, community-level intervention for MSM ages 15-25 (i.e., young MSM or YMSM). All 13 communities have some form of HIV-prevention activities naturally occurring in their jurisdiction, but 6 of the 13 communities were randomly assigned to also receive the multi-component intervention (1 additional city served as a case study and also received the intervention). This intervention includes 4 components: 1) community health advisor network (CHAN) consisting of YMSM who conduct outreach to their peers, including linking other YMSM to community services and conducting other parts of the intervention; 2) social marketing, to include the use media to disseminate HIV risk-reduction messages and promote positive norms for safer sex; 3) large group events with an HIV prevention theme; and 4) small group activities/workshops that focus on increasing HIV prevention skills and enhancing a positive self-identity.

The study population varies by site based on the specific racial or ethnic groups of YMSM that are targeted. African-American YMSM are the study population in Atlanta, Georgia (comparison site); Birmingham, Alabama (intervention site); and Chicago, Illinois (intervention site). Hispanic/Latino YMSM are the study population in Washington Heights/South Bronx, New York (intervention site); Jackson Heights/Queens, New York (comparison site); Orange County, California (intervention site); and San Gabriel Valley, California (comparison site). Asian and Pacific Islander YMSM are the study population in Seattle, Washington (intervention site) and San Diego, California (comparison site). YMSM regardless or race/ethnicity are the study population in Milwaukee, Wisconsin (intervention site); Detroit, Michigan (comparison site), Minneapolis, Minnesota (comparison site); and West Hollywood, California (intervention site).

The primary goals of the intervention are to 1) decrease UAI with any male partners; 2) decrease UAI with main male partners; and 3) decrease UAI with non-main (i.e., casual) male partners. Using a venue-based, time/space sampling strategy in each community, cross-sectional samples of YMSM were interviewed from May-August across 4 years (1999-2002). Data collected in 1999 and 2000 were prior to the implementation of the multi-component intervention, and data collected in 2001 and 2002 were during the implementation of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 15-25 years of age
* reports having sexual contact with another man in the past year
* meets the race/ethnicity eligibility criteria for the particular community

Exclusion Criteria:

Ages: 15 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12000
Dates: Start 1996-10; Primary Completion 2002-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
1) unprotected anal intercourse with a male partner in the past 3 months
2) unprotected anal intercourse at last sex with a main male partner (among participants with a male sex partner in the past 3 months and in the past year)
3) unprotected anal intercourse at last sex with the most recent non-main male partner (among participants with a male sex partner in the past 3 months and in the past year)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn A Guenther-Grey, M.A., Principal Investigator — Centers for Disease Control and Prevention
Locations (8):
- United States (8):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Childrens Hospital Los Angeles, Los Angeles, California
  - University of California-San Francisco, Center for AIDS Prevention Studies, San Francisco, California
  - Georgia State University, Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Education Development Center, Newton, Massachusetts
  - University of Minnesota Youth and AIDS Projects, Minneapolis, Minnesota
  - Medical College of Wisconsin, Center for AIDS Intervention Research, Milwaukee, Wisconsin

REFERENCES:
- [Background] Agronick G, O'Donnell L, Stueve A, Doval AS, Duran R, Vargo S. Sexual behaviors and risks among bisexually- and gay-identified young Latino men. AIDS Behav. 2004 Jun;8(2):185-97. doi: 10.1023/B:AIBE.0000030249.11679.d0. PMID 15187480
- [Background] Choi KH, Yep GA, Kumekawa E. HIV prevention among Asian and Pacific Islander American men who have sex with men: a critical review of theoretical models and directions for future research. AIDS Educ Prev. 1998 Jun;10(3 Suppl):19-30. PMID 9642428
- [Background] Choi KH, Kumekawa E, Dang Q, Kegeles SM, Hays RB, Stall R. Risk and protective factors affecting sexual behavior among young Asian and Pacific Islander men who have sex with men: Implications for HIV prevention. Journal of Sex Education and Therapy, 24(1&2): 47-55, 1999.
- [Background] Choi KH, Han CS, Hudes ES, Kegeles S. Unprotected sex and associated risk factors among young Asian and Pacific Islander men who have sex with men. AIDS Educ Prev. 2002 Dec;14(6):472-81. doi: 10.1521/aeap.14.8.472.24114. PMID 12512848
- [Background] Guenther-Grey CA, Varnell S, Weiser JI, Mathy RM, O'Donnell L, Stueve A, Remafedi G; Community Intervention Trial for Youth Study Team. Trends in sexual risk-taking among urban young men who have sex with men, 1999-2002. J Natl Med Assoc. 2005 Jul;97(7 Suppl):38S-43S. PMID 16080456
- [Background] Hart T, Peterson JL; Community Intervention Trial for Youth Study Team. Predictors of risky sexual behavior among young African American men who have sex with men. Am J Public Health. 2004 Jul;94(7):1122-4. doi: 10.2105/ajph.94.7.1122. PMID 15226130
- [Background] Mashburn AJ, Peterson JL, Bakeman R, Miller RL, Clark LF, and the Community Intervention Trial for Youth Study Team. Influences on HIV testing among young African-American men who have sex with men and the moderating effect of the geographic setting. Journal of Community Psychology 32(1): 45-60, 2004.
- [Background] Miller RL, Bedney BJ, Guenther-Grey C; CITY Project Study Team. Assessing organizational capacity to deliver HIV prevention services collaboratively: tales from the field. Health Educ Behav. 2003 Oct;30(5):582-600. doi: 10.1177/1090198103255327. PMID 14582599
- [Background] Muhib FB, Lin LS, Stueve A, Miller RL, Ford WL, Johnson WD, Smith PJ; Community Intervention Trial for Youth Study Team. A venue-based method for sampling hard-to-reach populations. Public Health Rep. 2001;116 Suppl 1(Suppl 1):216-22. doi: 10.1093/phr/116.S1.216. PMID 11889287
- [Background] O'Donnell L, Agronick G, San Doval A, Duran R, Myint-U A, Stueve A. Ethnic and gay community attachments and sexual risk behaviors among urban Latino young men who have sex with men. AIDS Educ Prev. 2002 Dec;14(6):457-71. doi: 10.1521/aeap.14.8.457.24109. PMID 12512847
- [Background] Peterson JL, Bakeman R, Stokes J, and the Community Intervention Trial for Youth Study Team. Racial/ethnic patterns of HIV sexual risk behaviors among young men who have sex with men. Journal of the Gay and Lesbian Medical Association 5(4): 155-162, 2001.
- [Background] Remafedi G. Suicidality in a venue-based sample of young men who have sex with men. J Adolesc Health. 2002 Oct;31(4):305-10. doi: 10.1016/s1054-139x(02)00405-6. PMID 12359375
- [Background] Seal DW, Bloom FR, Somlai AM. Dilemmas in conducting qualitative sex research in applied field settings. Health Educ Behav. 2000 Feb;27(1):10-23. doi: 10.1177/109019810002700102. PMID 10709789
- [Background] Seal DW, Kelly JA, Bloom FR, Stevenson LY, Coley BI, Broyles LA. HIV prevention with young men who have sex with men: what young men themselves say is needed. Medical College of Wisconsin CITY Project Research Team. AIDS Care. 2000 Feb;12(1):5-26. doi: 10.1080/09540120047431. PMID 10716014
- [Background] Stueve A, O'Donnell LN, Duran R, San Doval A, Blome J. Time-space sampling in minority communities: results with young Latino men who have sex with men. Am J Public Health. 2001 Jun;91(6):922-6. doi: 10.2105/ajph.91.6.922. PMID 11392935
- [Background] Stueve A, O'Donnell L, Duran R, San Doval A, Geier J; Community Intervention Trial for Youth Study Team. Being high and taking sexual risks: findings from a multisite survey of urban young men who have sex with men. AIDS Educ Prev. 2002 Dec;14(6):482-95. doi: 10.1521/aeap.14.8.482.24108. PMID 12512849